CLINICAL TRIAL: NCT06946355
Title: Food-based Randomized Trial for Enhancing Support of Hospitalized Children and Their Families
Brief Title: Food-based Support for Hospitalized Children and Their Families
Acronym: FRESH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 2023-0331; 1R01HD114702-01A1 (NIH)
Record Dates: First submitted 2025-04-02; First posted 2025-04-27 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Food Insecurity
Keywords: Pediatric; Hospitalization; Food Intake

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard Care (No Intervention): No post-discharge food support offered; no in-hospital food support offered; social work consults available per standard of care
- Both In-Hosptial and Post-Discharge (Active Comparator): The study team will provide two meals to up to two parents per day (for a maximum of four meals per day) in the hospital. The study team will provide families with a grocery gift card and frozen meals at the time of discharge.
  Interventions: Other: In-hospital food support intervention; Other: Post-discharge food support intervention
- Post-Discharge No In-Hospital (Active Comparator): The study team will provide families with a grocery gift card and frozen meals at the time of discharge. No in-hospital food support offered; social work consults available per standard of care.
  Interventions: Other: Post-discharge food support intervention
- In-Hospital No Post-Discharge (Active Comparator): The study team will provide two meals to up to two parents per day (for a maximum of four meals per day) in the hospital. No post-discharge food support offered; social work consults available per standard of care.
  Interventions: Other: In-hospital food support intervention

INTERVENTIONS:
Other: In-hospital food support intervention — The in-hospital food support intervention will provide two meals for up to two parents per day.
  Arms: Both In-Hosptial and Post-Discharge; In-Hospital No Post-Discharge
Other: Post-discharge food support intervention — The post-discharge intervention will provide families with grocery gift cards and frozen meals at the time of discharge.
  Arms: Both In-Hosptial and Post-Discharge; Post-Discharge No In-Hospital

SUMMARY:
The goal of this clinical trial is to learn if an intervention to provide food support to families who are part of government or self-pay insurances will provide benefits. The main questions it aims to answer are:

* Determine the effect of implementing an in-hospital food support intervention for low-income parents on reutilization and family-centered outcomes.
* Among families with baseline food insecurity, determine the effectiveness of a post-discharge food support intervention and as-needed social work referral on reutilization and family-centered outcomes.

Researchers will compare the in-hospital food support intervention and will be rolled out to sequential hospital units. In addition, the post-discharge food support intervention will be compared to standard discharge.

Some participants will:

* Receive in-hospital meal cards or standard care during hospitalization
* Receive post-discharge food support intervention or standard discharge
* Complete a 14-day post discharge follow-up survey

ELIGIBILITY:
Inclusion Criteria:

* All families of patients less than 21 years of age with Medicaid insurance or uninsured will be eligible

Exclusion Criteria:

* Patients admitted for end-of-life care, patients who will be discharged to a location other than home, patients who live independently, and patients in county custody.

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9119 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day urgent reutilization | 30 days post-discharge
  Validated measure of unplanned readmission/ED/urgent care use via electronic health record (EHR)
Hunger during hospitalization | Within 36 hours before discharge
  USDA Six-Item Short Form of the Food Security Survey Module, adapted to measure hunger in hospital. Families with lower scores are less likely to experience food insecurity. The family's level of food insecurity increases with the score.
  * Raw score 0-1-High food security
  * Raw score 2-4-Low food security
  * Raw score 5-6-Very low food security
Post-discharge hunger and food insecurity | 14 Days post-discharge
  USDA Six-Item Short Form of the Food Security Survey Module. Families with lower scores are less likely to experience food insecurity. The family's level of food insecurity increases with the score.
  * Raw score 0-1-High food security
  * Raw score 2-4-Low food security
  * Raw score 5-6-Very low food security

SECONDARY OUTCOMES:
30-day unplanned readmission | 30 Days post-discharge
  Validated measure of unplanned readmission
30-day Emergency department utilization | 30 Days post-discharge
  Emergency department utilization
Understanding of discharge instructions Confidence in care at home | 14 Days post-discharge
  Pediatric Transition Experience Measure (P-TEM)-Transition Preparation Domain
Return to normal routine | 14 Days post-discharge
  Family designed measure that assesses a family's return to normal routines
Post-Discharge coping | 14 Days post-discharge
  Post-Discharge Difficulty Coping Scale is measured at 14-day post-discharge phone call. Post-Discharge Coping Difficulty Scale uses an 11-point scaling format (0-10) with total scores ranging from 0 to 100. Higher scores represent greater coping difficulty.
Out of pocket expenses | Within 36 hours before discharge
  Expenses paid by the family during the hospitalization
Ability to pay for medications | 14 Days post-discharge
  Family-reported measure regarding difficulty paying for medications

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Auger, Principal Investigator — katherine.auger@cchmc.org
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States